CLINICAL TRIAL: NCT07138963
Title: Phenotype - Genotype Correlation in a Sample of Egyptian Patients With Congenital Myopathies and Congenital Muscular Dystrophies
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nouran Mohamed Sabry Abdel Aziz, Assistant Lecturer of Neurology and Psychiatry Department, Faculty of Medicine, Ain Shams University, Egypt., Ain Shams University
Other Study IDs: FMASU MD103/2024
Record Dates: First submitted 2025-07-31; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Phenotype; Genotype; Correction; Sample; Egyptian Patients; Congenital Myopathies; Congenital Muscular Dystrophies
MeSH Terms: conditions — Myotonia Congenita | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Patients with congenital myopathies or congenital muscular dystrophies evaluated for phenotype-genotype correlation.
  Interventions: Diagnostic Test: Genetic Testing and Muscle Biopsy

INTERVENTIONS:
Diagnostic Test: Genetic Testing and Muscle Biopsy — Comprehensive diagnostic assessment including clinical examination, electromyography (EMG), muscle biopsy for histopathological evaluation, and genetic testing to determine phenotype-genotype correlation in congenital myopathies and muscular dystrophies.

SUMMARY:
The aim of this study is to correlate the phenotype and genotype among a sample of Egyptian patients with Congenital myopathies and Congenital muscular dystrophies.

DETAILED DESCRIPTION:
Congenital Muscular dystrophies (CMDs) and Congenital Myopathies (CMs) constitute the two most important groups of congenital muscle diseases with early onset whether at birth or early infancy.

CMDs and CMs as a group encompass great clinical and genetic heterogeneity so that achieving an accurate genetic diagnosis has become increasingly challenging, even in the era of next generation sequencing. However, it has become clear that there is overlap between CMDs and CMs on the clinical, pathological and genetic level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical criteria of Congenital Myopathies (CMs) and Congenital Muscular dystrophies (CMDs) with different modes of inheritance.
* Age: patients below age of 18 years.
* Gender: Both males and females are included
* Genetically confirmed CMs and CMDs.

Exclusion Criteria:

* Patients above 18 years.
* Spinal muscular atrophy (SMA),and root lesions.
* Congenital myasthenic syndromes
* Dystrophinopathies,Duchenne Muscular Dystrophy (DMD), Limb-Girdle Muscular Dystrophy (LGMD)
* .Metabolic myopathies
* .Inflammatory muscle diseases

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Descriptive Cross-sectional study was caried out on patients with suspected or confirmed congenital myopathies or congenital muscular dystrophies presenting to Ain Shams University Hospitals, recruited over a specific study period.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Phenotype and genotype of congenital myopathies (CM) and congenital muscular dystrophies (CMD) patients | Two years
  Correlation of the most common clinical presentations and complications among Egyptian patients with congenital myopathies (CM) and congenital muscular dystrophies (CMD) of different genotypes.

SECONDARY OUTCOMES:
Common facial features | Two years
  Identification and comparison of typical dysmorphic facial features associated with different genetic subtypes of congenital myopathies (CM) and congenital muscular dystrophies (CMD).
Response to physiotherapy | Two years
  Response to physiotherapy will be recorded.
Prognosis of same genotype across different age groups | Two years
  The prognosis of the same genotype across different age groups will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author